CLINICAL TRIAL: NCT00393861
Title: Phase II Study of Oxaliplatin Plus Bevacizumab Salvage Chemotherapy in Patients With Germ Cell Tumors
Brief Title: Study of Oxaliplatin Plus Bevacizumab in Germ Cell Tumor Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0609-11; IUCRO-0166; IUCRO-0166 (Other: Indiana Univesity Simon Cancer Center); AVF4003s (Other: Industry Drug Sponsor)
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Neoplasms, Germ Cell and Embryonal
Keywords: Germ Cell Tumor; Germ Cell Cancer
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal | interventions — Bevacizumab; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oxaliplatin & bevacizumab (Experimental)
  Interventions: Drug: Bevacizumab and Oxaliplatin

INTERVENTIONS:
Drug: Bevacizumab and Oxaliplatin — Oxaliplatin 85 mg/M2 IV over 2 hours plus Bevacizumab 10 mg/kg IV over 90 minutes

SUMMARY:
The purpose of this study is to evaluate the effectiveness of oxaliplatin and bevacizumab in patients with refractory or relapsed germ cell tumors.

DETAILED DESCRIPTION:
This study proposes to look at the established combination of oxaliplatin and bevacizumab as used in colorectal cancer in refractory germ cell tumor patients. Oxaliplatin is a drug of known activity. Although bevacizumab has no single agent data, it combines dramatically well with numerous chemotherapy drugs, such as oxaliplatin increasing response rates and improving survival. Furthermore, VEG-F appears to be an important target in germ cell tumors as it does in so many other types of solid tumors. We will be using the identical dosages of oxaliplatin + bevacizumab as has been utilized in previously treated colorectal cancer, without the addition of 5-FU + leucovorin. This dose and schedule has been proven to be safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or serologic proof of metastatic germ cell neoplasm (gonadal or extragonadal primary). Patients with seminoma and non-seminoma are eligible, as are women with ovarian germ cell tumors.
* Patient's disease must not be amenable to cure with either surgery or chemotherapy in the opinion of the investigator.
* Patients must have failed initial cisplatin combination chemotherapy administered with curative intent such as BEP, EP, VIP, or similar regimens.
* Patients should have failed and demonstrated progressive disease with high dose chemotherapy such as carboplatin and etoposide. (With the exception of late relapse or primary mediastinal non-seminomatous germ cell tumor.
* Patients with late relapse or primary mediastinal non-seminomatous germ cell tumors must have failed at least 1 salvage chemotherapy regimen.
* Patients must have had prior exposure to paclitaxel, gemcitabine, or the combination of paclitaxel + gemcitabine.
* Patients must have adequate hematologic function (WBC > 4,000/mm3 and platelets > 100,000/mm3) obtained < 4 weeks prior to registration.
* Patients must have adequate hepatocellular function (SGOT < 4 x normal and Bilirubin <2.0 mg/dl) obtained < 4 weeks from protocol registration.
* Serum Creatinine must be < 2.0 mg/dl obtained < 4 weeks from protocol registration.
* Patients must have an ECOG performance status of 0, 1, or 2.
* Patients must be at least 28 days post major surgery, open biopsy, or significant traumatic injury at time of study registration.
* Patients must be at least 7 days post any minor surgical procedure, excluding placement of a vascular access device at the time of study registration.
* Patients must be at least 18 years old at time of consent.

Exclusion Criteria:

* Patients who have an active, unresolved infection and/or are receiving concurrent treatment with parenteral antibiotics are ineligible. Patients are eligible after antibiotics have been discontinued for at least 7 days.
* Patients may not have any significant bleeding.
* Patients with INR > 1.5 are not eligible unless the patient is on anti-coagulants with a therapeutic INR between 1.5 and 3. Patients on coumadin are not eligible unless they are on low dose coumadin to keep a vascular access device patent.
* Patients with a history of arterial thromboses, unstable angina, transient ischemic attach (TIA), cerebral vascular accident (CVA), or a myocardial infarction within the last 6 months are not eligible.
* Patients must not have known CNS metastases. A Head CT or MRI will be performed only if clinically indicated.
* Patients must not have received any radiotherapy or chemotherapy within 28 days prior to study registration, and have recovered from all toxicity from prior treatments.
* Patients must not have any prior history of hypertensive crisis or hypertensive encephalopathy.
* Patients must not have New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* Patients must not have history of significant vascular disease.
* Patients must not have evidence of bleeding diathesis or coagulopathy.
* Patients must not have inadequately controlled hypertension (defined as systolic blood pressure 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
* Patients must not have history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study registration.
* Patients must not have serious, non-healing would, ulcer or bone fracture.
* Patients must not have proteinuria at screening as demonstrated by a urine protein: Creatinine (UPC) ratio of ≥ 1.0.
* Patients must not have a known sensitivity to any component of bevacizumab.
* Patients must not be pregnant or lactating.
* Patients must not have grade 3 or 4 neuropathy.
* Females of child bearing potential must not be pregnant. A negative pregnancy test is required within 7 days prior to beginning treatment.

NOTE THE FOLLOWING GUIDELINES FOR USE IN THIS PROTOCOL:

* Progressive metastatic disease will be documented by the appearance of metastatic lesions on PA and lateral chest x-ray, C.T. scan, or other imaging studies, or the presence of a rising serum HCG or AFP.
* If a rising serum marker is the only evidence of progressive disease, at least 2 consecutive determinations must be done exhibiting serologic progression and alternative causes for increased serum levels of these substances must not be present [cross reaction with LH (tested if necessary by testosterone suppression of LH), ingestion of marijuana, hepatitis, etc.].
* Patients will be considered to have failed a prior regimen if they fail to obtain a complete response per RECIST as outlined in section 6.
* Patients with clinical situation of growing teratoma (normal or declining markers and radiographic or clinical progression) should be considered for surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-10; Primary Completion 2012-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Einhorn, MD, Principal Investigator — Indiana Univeristy School of Medicine
Locations (2):
- United States (2):
  - Indiana Univeristy Cancer Center, Indianapolis, Indiana
  - University of Pennsylvania:Abramson Cancer Center, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This protocol was based on getting at least 18 evaluable patients. Since the response data had looked promising, an additional 11 patients were added to obtain more accurate estimates of response.
Period: Overall Study
Arm/Group | Oxaliplatin & Bevacizumab
Started | 29
Completed | 3
Not Completed | 26
Not completed — Adverse Event | 2
Not completed — Disease Progression | 24

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (12.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Twelve Month Disease-free Survival Rate
Description: The percent of patients being disease-free at 12 months after treatment initiation will be estimated with a 90% exact binomial confidence interval for the percent of patients receiving drug.
Time Frame: 12 month post completion of treatment
Population: All patients enrolled and received treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 29
percentage of participants | 3.5 [0.2 to 15.3]

2. Secondary Outcome: Objective Response Rate (Complete and Partial Response)
Description: The percent of patients having an objective response (complete or partial response) will be estimated with a 90% exact binomial confidence interval for the percent of patients receiving drug per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: completion of study, up to 5 years
Population: All patients enrolled and received treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 29
percentage of participants | 27.6 [14.5 to 44.3]

3. Secondary Outcome: Duration of Remission (CR + PR)
Description: Will be examined using Kaplan-Meier estimates. Time from earliest confirmed remission criteria until death or progression will be calculated. If a patient continued to be in remission at the end of the study, they will be censored at their last evaluation in the analysis.
Time Frame: completion of study, up to 5 years
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 29
months | 4.7 [2.1 to 17.2]

4. Secondary Outcome: Overall Survival
Description: Will be examined using Kaplan-Meier estimates. Time until death or last evaluation will be calculated. If a patient did not die, they will be censored in the analysis.
Time Frame: completion of study, up to 5 years
Population: All patients enrolled and received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Oxaliplatin & Bevacizumab
Number analyzed (Participants) | 29
months | 7.7 [5.4 to 13.4]

ADVERSE EVENTS:
Time Frame: beginning of treatment until the end of the study for up to 5 years
Arm/Group | Oxaliplatin & Bevacizumab
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 15/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxaliplatin & Bevacizumab (N=29)
CONSTIPATION (Gastrointestinal disorders) | 4
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 3
NAUSEA (Gastrointestinal disorders) | 12
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 4
VOMITING (Gastrointestinal disorders) | 7
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 10
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2
INJECTION SITE REACTION/EXTRAVASATION CHANGES (General disorders) | 2
PAIN - OTHER (General disorders) | 4
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Respiratory, thoracic and mediastinal disorders) | 2
ANOREXIA (Metabolism and nutrition disorders) | 4
DIZZINESS (Nervous system disorders) | 2
INSOMNIA (Nervous system disorders) | 3
NEUROPATHY: SENSORY (Nervous system disorders) | 10
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 2
PAIN - HEAD/HEADACHE (General disorders) | 2
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 3
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 2
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 2
HYPERTENSION (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes